CLINICAL TRIAL: NCT03259971
Title: The Role of Probiotics PS128 in Movement Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201703061MIPA
Record Dates: First submitted 2017-08-16; First posted 2017-08-24 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-04

CONDITIONS: Rett Syndrome; Tourette Syndrome; Tic Disorders
Keywords: Rett syndrome; Tourette syndrome; Probiotic
MeSH Terms: conditions — Rett Syndrome; Tourette Syndrome; Tic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized double blind placebo-controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (for tic disorder) (Placebo Comparator): The placebo will be dispensed to equal the volume of 1 tablet of Probiotic PS128, which is taken orally in 2 divided doses, 12 hours apart during the study period of 2 months for Tic disorders.
  Interventions: Dietary Supplement: Placebo
- PS128 (tic disorder) (Active Comparator): The Probiotic group in tic disorder will take Probiotic-Lactobacillus plantarum PS128, which contain 300mg (3x10^10 CFU) Lactobacillus plantarum PS128 and 100mg of Microcrystalline Cellulose in each tablet. It will be taken orally in 2 divided doses, 12 hours apart during the study period of 2 months for Tic disorders.
  Interventions: Dietary Supplement: Probiotic-Lactobacillus plantarum PS128
- Placebo (for Rett syndrome) (Placebo Comparator): The placebo will be dispensed to equal the volume of 1 tablet of Probiotic PS128, which is taken orally in 2 divided doses, 12 hours apart during the study period of 4 months for Rett syndrome
  Interventions: Dietary Supplement: Placebo
- PS128 (Rett syndrome) (Active Comparator): The Probiotic group will take Probiotic-Lactobacillus plantarum PS128, which contain 300mg (3x10^10 CFU) Lactobacillus plantarum PS128 and 100mg of Microcrystalline Cellulose in each tablet. It will be taken orally in 2 divided doses, 12 hours apart during the study period of 4 months for Rett Syndrome.
  Interventions: Dietary Supplement: Probiotic-Lactobacillus plantarum PS128

INTERVENTIONS:
Dietary Supplement: Probiotic-Lactobacillus plantarum PS128 — Probiotic supplement of Lactobacillus plantarum PS128 , 1 tablet , twice a day , 12 hrs apart, lasting 2 months for Tic disorders and 4 months for Rett syndrome
  Other Names: Lactobacillus plantarum PS128
  Arms: PS128 (Rett syndrome); PS128 (tic disorder)
Dietary Supplement: Placebo — placebo , 1 tablet , twice a day , 12 hrs apart, lasting 2 months for Tic disorders and 4 months for Rett syndrome
  Arms: Placebo (for Rett syndrome); Placebo (for tic disorder)

SUMMARY:
Pediatric movement disorders comprise of a large number of different neurological diseases including Rett syndrome (RTT) and Tourette syndrome. Studies in the literature as well as our preliminary reports showed that Rett syndrome and Tourette syndrome/Tic disorders are associated with a dysbiosis of the gut microbiota compared to normal control. Probiotic Lactobacillus plantarum PS128 is a diet supplement that available for human consumption. Probiotic Lactobacillus plantarum PS128 had showed psychotropic effects such as ameliorate anxiety- and depression-like behaviors as well as altered the level of neurotransmitters such as dopamine in the brain in animal models, which might be through microbiota-gut-brain axis. Therefore, the purpose of this study is to access the possible neurobehavior effects of Probiotic Lactobacillus plantarum PS128 in Rett syndrome and Tic disorders/Tourette syndrome.

DETAILED DESCRIPTION:
The study is a placebo-controlled double-blind randomized study, to determine the benefits of probiotic Lactobacillus plantarum PS128 vs placebo on symptoms for Tic disorders; and the symptoms, behavior, or cognition for Rett syndrome.

Patients with the Rett syndrome and Tic disorders/Tourette syndrome will be recruited into our study.The study period will last 4 months for Rett syndrome patients, age one year-50years; while 2 months for Tic disorders/Tourette syndrome patient, age 5 years-18 years.

The study will be performed in National Taiwan University Children Hospital. The patients will have neuropsychological and gut microbiota evaluation before and at the end of the study. There will also be interim follow up evaluations each month after the patient start taking the probiotic or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Rett syndrome:
* Males and females who have classic or atypical RTT diagnosed under consensus criteria
* Age: 1-50 years
* Tic disorders:
* males and females with clinical diagnosis
* Age: 8-18years
* Treatment naive 4 weeks prior to study
* Those with standard medications, dosage stable 4 weeks prior to study
* AADC syndrome:
* Males and females with AADC diagnosis
* Age: 1-50 years

Exclusion Criteria:

* Those who took probiotic or probiotic related product 4 weeks prior to the study or during the study
* Those who took antibiotic 4 weeks prior to the study
* Those showing poor compliance with any aspect of the study
* Those had adverse reactions to PS128

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2017-08-25 (Actual); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-08-20 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological test (Mullen Scales of Early Learning) | Change at four months from baseline
  for Rett syndrome
Yale Global Tic Severity Scale (YGTSS) | Change at 2 months from baseline
  for Tic disorders

SECONDARY OUTCOMES:
RTT severity score | Change at four months from baseline
  For Rett syndrome
Dystonia status (Fahn Marsden rating scale/Unified Dystonia Rating Scale ) | Visit 1, Visit 2, Visit 3, Visit 4 (Up to 4 months)
  For Rett syndrome
Anxiety, Depression, and Mood Scale (ADAMS) | Change at four months from baseline
  For Rett syndrome
Ghuman-Folstein Screen for Social Interaction (SSI) | Change at four months from baseline
  For Rett syndrome
Vineland Adaptive Behavioral scale | Change at four months from baseline
  For Rett syndrome
Early social communication scales | Change at four months from baseline
  For Rett syndrome
Pediatric Evaluation of Disability Inventory | Change at four months from baseline
  For Rett syndrome
Stool and gut microbiota evaluation | Change at four months from baseline
  For Rett and Tic disorders
Child Behavior Checklist (CBCL) | Change at 2 months from baseline
  For Tic disorders
Continuous performance test | Change at 2 months from baseline
  For Tic disorders
The Migraine Disability Assessment Test | Change at 2 months from baseline
  For Tic disorders
Children's Depression Inventory | Change at 2 months from baseline
  For Tic disorders
Obsessive-compulsive inventory | Change at 2 months from baseline
  For Tic disorders
Swanson, Nolan and Pehlam version IV | Change at 2 months from baseline
  For Tic disorders

CONTACTS AND LOCATIONS:
Overall Officials: Wang-Tso Lee, MD,PhD, Principal Investigator — National Taiwan University Children Hospital
Locations (1):
- National Taiwan University Children Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong LC, Hsu CJ, Wu YT, Chu HF, Lin JH, Wang HP, Hu SC, Tsai YC, Tsai WC, Lee WT. Investigating the impact of probiotic on neurological outcomes in Rett syndrome: A randomized, double-blind, and placebo-controlled pilot study. Autism. 2024 Sep;28(9):2267-2281. doi: 10.1177/13623613231225899. Epub 2024 Feb 15. PMID 38361371